CLINICAL TRIAL: NCT03559738
Title: Comparative Study of Extracorporeal Shock Wave Lithotripsy and Ureteroscopy in Management of Upper Third Ureteral Calculi
Brief Title: ESWL vs URS in Management of Upper Third Ureteric Calculi
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Atef Abdelaziz Mostafa, Resident, Assiut University
Other Study IDs: ureteric stones
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Ureteral Stones

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients With Upper Ureteric Stones: Patients with upper ureteral stones more than 1cm and 1000 HU

SUMMARY:
comparative study of two treatment modalities (ureteroscopy and extracorporeal shock wave lithotripsy) in management of upper third ureteral calculi

DETAILED DESCRIPTION:
Large impacted upper ureteral calculus is defined as a stone located above the lower border of the fourth lumbar vertebra, remaining fixed at the same site for at least six weeks. Moreover, it is associated with hydronephrosis and/or prevents contrast medium from passing below the calculus on intravenous urography (IVU).Moreover, there is inability to pass a guidewire or catheter beyond the stone at initial attempts. The treatment for patients with large impacted proximal ureteral stone remains controversial; the surgical options for the treatment of proximal ureteral stones include extracorporeal shockwave lithotripsy (ESWL), Ureteroscopy, PCNL and rarely Laparoscopic or Open surgery. Every technique has its own limitations. The aim of this study is to compare and to evaluate the outcome and complications of two main treatments procedures for impacted proximal ureteral calculi, Extracorporeal Shock Wave Lithotripsy (ESWL) and Ureteroscopy.

Extracorporeal Shock Wave Lithotripsy (ESWL) and Ureteroscopy are two common modalities in the management of Proximal Ureteral Calculi.European Association of Urology (EAU) and American Urological Association (AUA) guidelines have recommended URS or ESWL as first-line treatment Options.ESWL is an effective and non-invasive treatment method in urolithiasis, particularly in stones located in the upper third of the ureters.However, URS is a more invasive technique when compared to ESWL, URS became the most efficient treatment method in proximal ureteral calculi after the development of small-caliber, semi-rigid and flexible endoscopes and the holmium:YAG laser. Today, the greatest dilemma faced by Urologists is to choose between ESWL and URS. A number of factors influence the final results of ESWLand if no fragmentation occurs after several unsuccessful sessions, the stone is considered ESWL-resistant; the case is deemed an ESWL-failure and the patient therefore undergoes URS.URS has been described as a salvage or second line treatment option in cases of ESWL-resistant calculi

ELIGIBILITY:
Inclusion Criteria:

- The study will include patients in the age group of 18-70 years with body mass index of less than or equal to 30 kg/m2 with Upper Ureteral Calculi more than or equal to 1 cm with density about 900 - 1100 HU

Exclusion Criteria:

* Patients with distal obstruction
* Impacted stones : An impacted stone is defined as a stone where a guidewire will not pass without ancillary measures and/or a stone that does not move when forceful irrigation is applied ureteroscopically
* Marked hydronephrosis : gross dilation/ballooning of the renal pelvis and calyces with loss of borders between the renal pelvis and calyces and renal atrophy seen as cortical thinning
* Radiolucent stones
* Pregnancy
* Stones in Children
* Spinal deformity
* Morbid obesity
* Patients on Aspirin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 60 cases will be assigned to either ESWL or URS randomly
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
identify best management for upper third ureter stones | 2 years
  Matched Pair Analysis of Extracorporeal Shock Wave Lithotripsy versus Ureteroscopy for the management of Upper Ureteral Calculi with relatively small study group by comparing like-for-like Stones